CLINICAL TRIAL: NCT00404274
Title: An Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Steady-State Warfarin When Co-administered With Repeat Doses of Casopitant [GW679769] in Healthy Adult Subjects.
Brief Title: A Study Testing the Effect and Safety of Casopitant (GW679769) While Taking Warfarin in Healthy Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NKV105097
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Nausea and Vomiting, Chemotherapy-Induced
Keywords: healthy human volunteer; GW679769; warfarin; casopitant
MeSH Terms: conditions — Nausea; Vomiting | interventions — casopitant; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment regimen A (Experimental): In treatment regimen A subject will co-administer casopitant and warfarin over three-day period (Day 1 150 milligram per day [mg/day], Day 2 50 mg/day, Day 3 50 mg/day) and from Days 4 to 10 subject will administer only warfarin.
  Interventions: Drug: Casopitant (GW679769) oral tablets; Drug: Warfarin oral tablets
- Treatment regimen B (Experimental): In treatment regimen B subject will co-administer casopitant 60 mg/day and warfarin for 14 days.
  Interventions: Drug: Casopitant (GW679769) oral tablets; Drug: Warfarin oral tablets
- Treatment regimen C (Experimental): In treatment regimen C subject will co-administer warfarin and casopitant 30 mg/day for 14 days.
  Interventions: Drug: Casopitant (GW679769) oral tablets; Drug: Warfarin oral tablets

INTERVENTIONS:
Drug: Casopitant (GW679769) oral tablets — Casopitant will be available in the dose strength of 20,30 or 50 mg
Drug: Warfarin oral tablets — Warfarin will be available in the dose strength of 5 mg
  Other Names: Casopitant (GW679769) oral tablets

SUMMARY:
GW679769 may affect liver enzymes that metabolize warfarin. This study is designed to test the extent of the GW679769 affect on Warfarin levels in humans.

ELIGIBILITY:
Inclusion criteria:

* Healthy subjects
* non-smoking
* Females cannot be able to have children
* Must be able to swallow and retain oral medication
* Understand and sign the written consent
* comply with the requirements and restrictions involved in an overnight 30 day confinement in a healthcare setting

Exclusion criteria:

* cannot participate if subject has a clinically relevant abnormality, medical condition, or circumstance that makes them unsuitable for the study per the study doctor.
* blood donation in excess of 1 pint within 56 days before dosing of medication
* iron deficiency
* history of drug or alcohol abuse or dependency within the past 6 months
* subjects cannot use any nicotine-containing products within the last 6 months
* positive for HIV, Hepatitis B or C
* use of prescription or non-prescription drug(s), herbal or dietary supplements or vitamins with 14 days prior to first dose of study medication
* consumption of any food or drink containing grapefruit, Seville oranges, kumquats, pomelos (or their juices) within 7 days of the first dose of study medication
* history of bleeding disorders or excessive bleeding
* female who has a positive pregnancy test
* female who is lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2007-03-18 (Actual); Study Completion 2007-03-18 (Actual)

PRIMARY OUTCOMES:
Plasma levels of Warfarin at Period 1: Day 9 to 14, Period 2: Day 2 & 3 and Day 5 to 16. | Period 1: Day 9 to 14, Period 2: Day 2 & 3 and Day 5 to 16.
Plasma levels of casopitant at Period 2: Day 2 & 3 and Day 5 to 16. | Period 2: Day 2 & 3 and Day 5 to 16.

SECONDARY OUTCOMES:
Clinical lab tests monitoring of International Normalized Ratio (INR) adverse events vital signs 12 lead ECGs liver function tests | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Buffalo, New York

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Kirby LC, Johnson BM, Adams LM, Eberwein DJ, Zhang K, Murray SC, Lates CD, Blum RA, Morris SR. Effect of casopitant, a novel NK-1 receptor antagonist, on the pharmacokinetics and pharmacodynamics of steady-state warfarin. J Clin Pharmacol. 2010 May;50(5):566-75. doi: 10.1177/0091270009346965. Epub 2010 Mar 10. PMID 20220045
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study NKV105097 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/NKV105097?search=study&search_terms=NKV105097#rs
- Available data/document: Individual Participant Data Set: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKV105097 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register